CLINICAL TRIAL: NCT04635839
Title: Randomized Control Trial of Unfractionated Heparin Thromboprophylaxis Dosing for Antepartum Hospitalizations
Brief Title: Heparin Prophylaxis Dosing for Antepartum Hospitalizations (HEPDOSE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Thalia Wong, MD, Co-Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-001799
Record Dates: First submitted 2020-11-09; First posted 2020-11-19 (Actual); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy Related; Antepartum DVT
Keywords: Thromboprophylaxis; Antepartum admission; Heparin
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Dosing (Active Comparator): Standard dose of unfractionated heparin
  Interventions: Drug: Standard Dose of Unfractionated Heparin
- Gestational Age-Based Dosing (Active Comparator): Dose of unfractionated heparin based on trimester of pregnancy
  Interventions: Drug: Gestational Age-Based Dose of Unfractionated Heparin

INTERVENTIONS:
Drug: Standard Dose of Unfractionated Heparin — 5,000 units subcutaneous unfractionated heparin every 12 hours
  Arms: Standard Dosing
Drug: Gestational Age-Based Dose of Unfractionated Heparin — * First trimester (< 14 weeks of gestation): 5,000 units subcutaneous unfractionated heparin every 12 hours
  * Second trimester (14-28 weeks of gestation): 7,500 units subcutaneous unfractionated heparin every 12 hours
  * Third trimester (> 28 weeks of gestation): 10,000 units subcutaneous unfractionated heparin every 12 hours
  Arms: Gestational Age-Based Dosing

SUMMARY:
This study is a randomized control trial to compare gestational age-based dosing with standard dosing of unfractionated heparin for thromboprophylaxis of hospitalized antepartum patients. The investigators aim to determine the effect of dosing on receipt of neuraxial anesthesia and pregnancy outcomes and evaluate the pharmacokinetics and pharmacodynamics of unfractionated heparin in pregnancy.

DETAILED DESCRIPTION:
Venous thromboembolism is one of the leading causes of maternal morbidity and mortality, and antepartum hospitalizations place pregnant patients at an even higher risk of developing thromboembolism. As a result, there is an increased emphasis on administering pharmacologic thromboprophylaxis for antepartum patients with prolonged hospitalizations. Previously, standard dosing of unfractionated heparin was widely adopted for thromboprophylaxis in the pregnant population. However, due to a suspected altered metabolism of unfractionated heparin in pregnancy resulting in a decrease response, the American College of Obstetricians and Gynecologists (ACOG) currently recommends considering gestational age-based dosing for unfractionated heparin for thromboprophylaxis in pregnancy with standard dosing as an alternative option. The data supporting altered dosing is very limited. In addition, increased dosing of heparin may result in challenges in anesthetic management, potentially limiting the receipt of neuraxial anesthesia resulting in increased need for general anesthesia associated with both increased maternal and fetal risks. The potential effects of higher prophylactic unfractionated heparin dosing in pregnant patients need to be further explored before being widely adopted for inpatient antepartum thromboprophylaxis. The investigators propose this study to provide a direct comparison of gestational age-based unfractionated heparin dosing to standard dosing of unfractionated heparin for pharmacologic thromboprophylaxis of hospitalized antepartum patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Speak English or Spanish
* Antepartum admission for at least 72 hours at Ronald Reagan UCLA Medical Center
* Provides informed consent for study participation

Exclusion Criteria:

* Active or threatened antenatal bleeding
* Disseminated intravascular coagulation
* Risk of imminent delivery (delivery within 12 hours)
* Thrombocytopenia (platelet count < 100 x 109)
* Elevated baseline aPTT (> 36.2 seconds)
* Concern for hemolysis, elevated liver enzymes, low platelet count (HELLP) syndrome
* Congenital bleeding disorders (hemophilias)
* Receiving therapeutic or prophylactic anticoagulation (unfractionated heparin, low molecular weight heparin, oral anticoagulants) for alternative indication (e.g., acquired or inherited thrombophilia, history of VTE)
* History of heparin-induced thrombocytopenia (HIT)
* SARS-CoV-2 positive
* Cognitive impairment, psychiatric instability, or language barriers that limit their ability to provide informed consent
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Mok T, Nguyen AV, Kwan L, Steinberg I, Vallera C, Silverman NS, Rao R. Prophylactic Unfractionated Heparin in Antepartum Hospitalizations: A Randomized Controlled Trial. Obstet Gynecol. 2024 Jul 1;144(1):118-125. doi: 10.1097/AOG.0000000000005599. Epub 2024 May 14. PMID 38743958

RESULTS

PARTICIPANT FLOW:
Groups:
- Gestational Age-Based Dosing: Dose of unfractionated heparin based on trimester of pregnancy
  Gestational Age-Based Dose of Unfractionated Heparin: - First trimester (< 14 weeks of gestation): 5,000 units subcutaneous unfractionated heparin every 12 hours
  * Second trimester (14-28 weeks of gestation): 7,500 units subcutaneous unfractionated heparin every 12 hours
  * Third trimester (> 28 weeks of gestation): 10,000 units subcutaneous unfractionated heparin every 12 hours
Period: Overall Study
Arm/Group | Standard Dosing | Gestational Age-Based Dosing
Started | 22 | 24
Completed | 21 | 24
Not Completed | 1 | 0
Not completed — Delivered prior to second dose of heparin | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dosing | Gestational Age-Based Dosing | Total
Number analyzed (Participants) | 21 | 24 | 45
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [28 to 36] | 34 [31 to 38] | 33 [28 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 12 | 21
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 5 | 11 | 16
  More than one race | 11 | 6 | 17
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 21 | 24 | 45
Gravida [Median (Inter-Quartile Range); unit: pregnancies] | 2 [1 to 3] | 2 [2 to 5] | 2 [1 to 3]
Nulliparous [Count of Participants; unit: Participants] | 15 | 10 | 25
Gestational age at randomization [Median (Inter-Quartile Range); unit: weeks] | 30.3 [26.4 to 32.6] | 30.4 [27.6 to 33.0] | 30.3 [27.1 to 32.6]
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 29.9 [27.6 to 33.2] | 30.4 [27.6 to 33.0] | 30.1 [27.4 to 33.1]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Elevated Serum Activated Partial Thromboplastin Time Above the Normal Range (> 36.2 Seconds).
Description: Surrogate marker for whether or not the patient would be eligible for neuraxial anesthesia based on guidelines for neuraxial anesthesia in pregnant women receiving VTE prophylaxis
Time Frame: Collected 6 hours after unfractionated heparin dose until patient was taken of unfractionated heparin, an average of 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dosing | Gestational Age-Based Dosing
Number analyzed (Participants) | 21 | 24
Participants | 1 | 8

2. Secondary Outcome: Number of Participants Diagnosed With Venous Thromboembolism (Pulmonary Embolism and/or Deep Venous Thromboembolism)
Time Frame: Assessed throughout hospitalization, an average length of 8 days, until 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dosing | Gestational Age-Based Dosing
Number analyzed (Participants) | 21 | 24
Participants | 1 | 0

3. Secondary Outcome: Number of Participants Who Did Not Receive or Had a Delay of Neuraxial Anesthesia Due to Unfractionated Heparin
Time Frame: Assessed at time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dosing | Gestational Age-Based Dosing
Number analyzed (Participants) | 21 | 24
Participants | 0 | 0

4. Secondary Outcome: Number of Participants That Received General Anesthesia
Time Frame: Assessed at time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dosing | Gestational Age-Based Dosing
Number analyzed (Participants) | 21 | 24
Participants | 1 | 0

5. Secondary Outcome: Number of Participants That Had a Delay in Timing of Delivery Due to Unfractionated Heparin
Time Frame: Assessed at time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dosing | Gestational Age-Based Dosing
Number analyzed (Participants) | 21 | 24
Participants | 0 | 0

6. Secondary Outcome: Maximum Anti-Factor Xa Level Measured
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: IU/mL
Arm/Group | Standard Dosing | Gestational Age-Based Dosing
Number analyzed (Participants) | 21 | 24
IU/mL | 0.09 [0.09 to 0.09] | 0.09 [0.09 to 0.11]

7. Secondary Outcome: Mode of Delivery
Time Frame: Assessed at time of delivery
Population: 1 participant in Arm 1 (standard dosing) delivered at an outside hospital and mode of delivery is unavailable
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dosing | Gestational Age-Based Dosing
Number analyzed (Participants) | 20 | 24
Participants
  Vaginal delivery | 6 | 4
  Cesarean delivery | 14 | 20

8. Secondary Outcome: Estimated Blood Loss From Delivery
Time Frame: Assessed at time of delivery
Population: 1 participant in Arm 1 (standard dosing) delivered at an outside hospital and estimated blood loss is unavailable
Measure: Median (Inter-Quartile Range); unit: cc
Arm/Group | Standard Dosing | Gestational Age-Based Dosing
Number analyzed (Participants) | 20 | 24
cc | 654 [125 to 1344] | 593 [505 to 905]

9. Secondary Outcome: Number of Participants That Received a Blood Transfusion
Time Frame: From time of delivery until 6 weeks after delivery
Population: 1 participant in Arm 1 (standard dosing) delivered at an outside hospital and need for blood transfusion is unavailable
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dosing | Gestational Age-Based Dosing
Number analyzed (Participants) | 20 | 24
Participants | 1 | 7

10. Secondary Outcome: Maximum Activated Partial Thromboplastin Clotting Time Levels Measured
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Standard Dosing | Gestational Age-Based Dosing
Number analyzed (Participants) | 21 | 24
seconds | 26.6 [23.0 to 29.6] | 30.4 [7.4 to 37.5]

ADVERSE EVENTS:
Time Frame: Adverse event data was evaluated and collected from time of enrollment in study until 6 weeks after study completion, an average of 8 weeks.
Description: Adverse events were routinely monitored and assessed for by the principal investigator through medical chart review.
Arm/Group | Standard Dosing | Gestational Age-Based Dosing
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/24
Other Adverse Events (participants affected / at risk) | 0/21 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT04635839/Prot_004.pdf
  • Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT04635839/SAP_005.pdf
  • Informed Consent Form (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT04635839/ICF_006.pdf